CLINICAL TRIAL: NCT01268605
Title: Resin Based Composite Occlusal Restoration Postoperative Hypersensitivity: Randomized Comparative Effectiveness Research Trial
Brief Title: Postoperative Hypersensitivity Randomized Comparative Effectiveness Research Trial
Acronym: POH RCERT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pearl Network (Network)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRL1013; U01DE016755 (NIH); 136277 (Other Grant/Funding Number: NIDCR)
Record Dates: First submitted 2010-10-19; First posted 2010-12-31 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Dental Caries
Keywords: Dental caries; Resin based composite; Hypersensitivity; Teeth; Dentistry; Practice-based research network
MeSH Terms: conditions — Dental Caries; Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Restoration with a dentin bonding agent (DBA) (Active Comparator): Restoration with a dentin bonding agent (DBA) and hybrid resin-based composite: Use of a self-etch DBA Clearfil SE Bond followed by Herculite Ultra resin-based composite (Sybron/Kerr), comprising a state-of-the-art bonding and restoration system for cervical lesions.
  Interventions: Procedure: Restoration with a dentin bonding agent (DBA)
- Restoration with a resin modified glass ionomer liner (RMGI) (Active Comparator): Restoration with a resin modified glass ionomer liner (RMGI) (Vitrebond LC, placed on the pulpal floor at a thickness of approximately 0.5 mm) followed by application of a two step self etch DBA and nanofilled resin based composite (RBC).
  Interventions: Procedure: Restoration with a resin modified glass ionomer liner (RMGI)

INTERVENTIONS:
Procedure: Restoration with a dentin bonding agent (DBA) — Restoration with a dentin bonding agent (DBA) and hybrid resin-based composite: Use of a self-etch DBA Clearfil SE Bond followed by Herculite Ultra resin-based composite (Sybron/Kerr), comprising a state-of-the-art bonding and restoration system for cervical lesions.
  Arms: Restoration with a dentin bonding agent (DBA)
Procedure: Restoration with a resin modified glass ionomer liner (RMGI) — Restoration with a resin modified glass ionomer liner (RMGI) (Vitrebond LC, placed on the pulpal floor at a thickness of approximately 0.5 mm) followed by application of a two step self etch DBA and nanofilled resin based composite (RBC).
  Arms: Restoration with a resin modified glass ionomer liner (RMGI)

SUMMARY:
Postoperative hypersensitivity (POH) is a problem for many patients as determined by the recent Practitioners Engaged in Applied Research and Learning (PEARL) study of POH following occlusal caries restoration. The objectives of this two-armed randomized comparative effectiveness research trial (RCERT) are to determine whether adding a resin modified glass ionomer liner (RMGI) reduces POH in dentin bonded Class I resin based composite (RBC) restorations, and to identify other factors (putative risk factors) that are associated with increased POH.

The primary outcome of this study is the reduction/elimination of restoration POH as measured by clinical assessment (air stream) and patient-reports.

Outcomes will be ascertained via the following specific aims:

Specific Aim 1: To compare the reduction of hypersensitivity of study teeth by clinical measurement (air drying) and by patient-reported outcomes among the two treatment groups at three points in time: prior to restoration and at one and four weeks postrestoration.

Specific Aim 2: To identify putative risk factors for POH (or factors associated with differences in POH) including: preoperative caries stage measured by the proposed American Dental Association (ADA) Caries Classification System (CCS), lesion depth as measured on the preoperative radiograph, dentin caries activity ranked on opening the lesion, preparation depth, and patient sleep bruxism status.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of solely adult dentition ages 15 to 60 (The upper age of 60 years is selected since the pulp space is limited and POH is less likely above this age).
2. Presence of one or more permanent posterior teeth (in different quadrants, with third molars excluded) with the clinical diagnosis of new Class I caries extending into dentin with or without radiographic confirmation. Up to 4 teeth (one per quadrant) may be enrolled. If there is more than one occlusal lesion in a quadrant that meets the inclusion criteria the patient is not eligible for inclusion in the study. Only one tooth per quadrant can be treated during the 4 weeks of this study.
3. Lesion depth, if visible on radiograph, must be ≤1/2 the distance from the Dento-Enamel Junction (DEJ) to the pulp and the radiograph cannot be more than 9 months old.
4. The tooth must be in occlusion with a natural tooth.
5. A resin-based composite restoration would be the standard of care for the lesion.
6. The tooth must be free of evidence of a pulpitis (no report of lingering pain associated with any stimulus).
7. Subjects must be available for contact for at least four weeks post-treatment.
8. Subjects willing and able to understand and sign the IRB-approved informed consent form and for individuals under the age of 18, the parental / guardian assent form.
9. Subject's baseline score on the NPAS must be ≥3 for air and/or cold stimulation but not exhibit pain lasting more than approximately four seconds which is known as "lingering pain"
10. Gingival Index of less than or equal to 2.

Exclusion Criteria:

1. Individuals in which the second molars are not fully erupted.
2. Teeth with a mobility of 2 or greater, or inflamed gingival tissues.
3. Existing restoration(s) on the same tooth.
4. Teeth that have been clinically assessed to be fractured.
5. Tooth is an abutment for a removable partial denture.
6. Tooth with subgingival calculus, unless removed during the treatment visit.
7. Subjects undergoing active orthodontic treatment. Use of retainers is allowed.
8. Subjects currently enrolled in or who have completed in the past month a tooth bleaching program.
9. Subjects with prior reaction or inability to tolerate any of the dental products being used, such as severe topical or hypersensitivity reaction.
10. Subjects under treatment for medical disorders including: dementia, Parkinson's disease, severe depression, severe anxiety, and any other medical condition that, in the opinion of the P-I, would affect the subject's judgment of postoperative hypersensitivity and ability to understand the informed consent process.
11. Subjects in another ongoing dental research study.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 341 (Actual)
Dates: Start 2010-09; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Hypersensitivity | 4 weeks
  To compare the reduction of hypersensitivity of study teeth by clinical measurement (air drying) and by patient-reported outcomes among the two treatment groups at three points in time: prior to restoration and at one and four weeks postrestoration.

SECONDARY OUTCOMES:
Preoperative caries stage | Baseline
  To identify putative risk factors for POH (or factors associated with differences in POH) including: preoperative caries stage measured by the proposed ADA Caries Classification System (CCS), lesion depth as measured on the preoperative radiograph, dentin caries activity ranked on opening the lesion, preparation depth, and patient sleep bruxism status.
Lesion depth | Baseline
  To identify putative risk factors for POH (or factors associated with differences in POH) including: preoperative caries stage measured by the proposed ADA Caries Classification System (CCS), lesion depth as measured on the preoperative radiograph, dentin caries activity ranked on opening the lesion, preparation depth, and patient sleep bruxism status.
Dentin caries activity | Baseline
  To identify putative risk factors for POH (or factors associated with differences in POH) including: preoperative caries stage measured by the proposed ADA Caries Classification System (CCS), lesion depth as measured on the preoperative radiograph, dentin caries activity ranked on opening the lesion, preparation depth, and patient sleep bruxism status.
Preparation depth | Baseline
  To identify putative risk factors for POH (or factors associated with differences in POH) including: preoperative caries stage measured by the proposed ADA Caries Classification System (CCS), lesion depth as measured on the preoperative radiograph, dentin caries activity ranked on opening the lesion, preparation depth, and patient sleep bruxism status.
Sleep bruxism status | Baseline
  To identify putative risk factors for POH (or factors associated with differences in POH) including: preoperative caries stage measured by the proposed ADA Caries Classification System (CCS), lesion depth as measured on the preoperative radiograph, dentin caries activity ranked on opening the lesion, preparation depth, and patient sleep bruxism status.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick A Curro, DMD, Phd, Principal Investigator — NYU Langone Health
Locations (41):
- United States (41):
  - Phoenix Pediatric Dental, Phoeniz, Arizona
  - Watson and Niven Dental Partnership, Newport Beach, California
  - Jana A. Ikeda, DDS, PC, Boulder, Colorado
  - Maryann Lehmann, D.D.S., Darien, Connecticut
  - Oracare Research, Sanford, Florida
  - Complete Dental Arts, P.C., Newnan, Georgia
  - Creative Smiles Dental Care, Champaign, Illinois
  - Peggy Richardson, DDS, MS, Tinley Park, Illinois
  - Kokomo Oral Implantology, Kokomo, Indiana
  - Corridor Kids Pediatric Dentistry, North Liberty, Iowa
  - Community Dental - Biddeford Center, Biddeford, Maine
  - Cheryl F, Callahan, DDS, PA, Rockville, Maryland
  - Oral Medicine - Tufts School of Dental Medicine, Boston, Massachusetts
  - Frank A Dahlstrom,DMD,PC, Dennis, Massachusetts
  - Oral Health Center, Southborough, Massachusetts
  - Small Smiles Dental Center of Springfield, LLC, Springfield, Massachusetts
  - Keith A Hudson DDS PC, Franklin, Michigan
  - Minnesota Dentalcare, Richfield, Minnesota
  - Eric Hirschfeld, D.D.S., Conway, New Hampshire
  - Bordentown Family Dental, Bordentown, New Jersey
  - Scott B Schaffer, DMD, Clark, New Jersey
  - Gentle Dental Care, LLC, Edison, New Jersey
  - Dr. Howard Spielman, Plainsboro, New Jersey
  - Barry G. Dale, DMD, Tenafly, New Jersey
  - Cynthia Jetter, DMD, Voorhees Township, New Jersey
  - Bay Dental PC, Brooklyn, New York
  - Eric Leibowitz DDS, Brooklyn, New York
  - Queens Comprehensive Dental Services, Forest Hills, New York
  - Gilberto Nunez DDS LLC, Kingston, New York
  - Kay T. Oen, DDS, Port Chester, New York
  - East Avenue Dentistry PLLC, Rochester, New York
  - James R. Keenan, DDS, PC, Rockaway Beach, New York
  - Janice K. Pliszczak, DDS, Syracuse, New York
  - Susan D. Bernstein, DDS, Cincinnati, Ohio
  - Laurence H Stone, DDS, Doylestown, Pennsylvania
  - Dr. Jeannette Abboud-Niemczyk, Drexel Hill, Pennsylvania
  - Allan J Horowitz, DMD, King of Prussia, Pennsylvania
  - Dr. Julie Ann Barna, Lewisburg, Pennsylvania
  - Salvation Army Dental Center, Oil City, Pennsylvania
  - Elizabeth W. Galloway, Hilton Head Island, South Carolina
  - MEHOP, Bay City, Texas

REFERENCES:
- [Background] American Academy of Sleep Medicine (2001). The international classification of sleep disorders, revised: diagnosis and coding manual. Westchester, IL: American Academy of Sleep Medicine.
- [Background] Akpata ES, Sadiq W. Post-operative sensitivity in glass-ionomer versus adhesive resin-lined posterior composites. Am J Dent. 2001 Feb;14(1):34-8. PMID 11806478
- [Background] Akpata ES, Behbehani J. Effect of bonding systems on post-operative sensitivity from posterior composites. Am J Dent. 2006 Jun;19(3):151-4. PMID 16838478
- [Background] Auschill TM, Koch CA, Wolkewitz M, Hellwig E, Arweiler NB. Occurrence and causing stimuli of postoperative sensitivity in composite restorations. Oper Dent. 2009 Jan-Feb;34(1):3-10. doi: 10.2341/08-7. PMID 19192831
- [Background] Baratieri LN, Ritter AV. Four-year clinical evaluation of posterior resin-based composite restorations placed using the total-etch technique. J Esthet Restor Dent. 2001;13(1):50-7. doi: 10.1111/j.1708-8240.2001.tb00251.x. PMID 11831309
- [Background] Briso AL, Mestrener SR, Delicio G, Sundfeld RH, Bedran-Russo AK, de Alexandre RS, Ambrosano GM. Clinical assessment of postoperative sensitivity in posterior composite restorations. Oper Dent. 2007 Sep-Oct;32(5):421-6. doi: 10.2341/06-141. PMID 17910217
- [Background] Browning WD, Blalock JS, Callan RS, Brackett WW, Schull GF, Davenport MB, Brackett MG. Postoperative sensitivity: a comparison of two bonding agents. Oper Dent. 2007 Mar-Apr;32(2):112-7. doi: 10.2341/06-58. PMID 17427818
- [Background] Casselli DS, Martins LR. Postoperative sensitivity in Class I composite resin restorations in vivo. J Adhes Dent. 2006 Feb;8(1):53-8. PMID 16536346
- [Background] Cho BH, Dickens SH, Bae JH, Chang CG, Son HH, Um CM. Effect of interfacial bond quality on the direction of polymerization shrinkage flow in resin composite restorations. Oper Dent. 2002 May-Jun;27(3):297-304. PMID 12022463
- [Background] Christensen GJ. Preventing postoperative tooth sensitivity in class I, II and V restorations. J Am Dent Assoc. 2002 Feb;133(2):229-31. doi: 10.14219/jada.archive.2002.0149. PMID 11868844
- [Background] Efes BG, Dorter C, Gomec Y, Koray F. Two-year clinical evaluation of ormocer and nanofill composite with and without a flowable liner. J Adhes Dent. 2006 Apr;8(2):119-26. PMID 16708724
- [Background] Ernst CP, Martin M, Stuff S, Willershausen B. Clinical performance of a packable resin composite for posterior teeth after 3 years. Clin Oral Investig. 2001 Sep;5(3):148-55. doi: 10.1007/s007840100117. PMID 11642558
- [Background] Ernst CP, Brandenbusch M, Meyer G, Canbek K, Gottschalk F, Willershausen B. Two-year clinical performance of a nanofiller vs a fine-particle hybrid resin composite. Clin Oral Investig. 2006 Jun;10(2):119-25. doi: 10.1007/s00784-006-0041-8. Epub 2006 Mar 23. PMID 16555069
- [Background] Gordan VV, Mjor IA. Short- and long-term clinical evaluation of post-operative sensitivity of a new resin-based restorative material and self-etching primer. Oper Dent. 2002 Nov-Dec;27(6):543-8. PMID 12413217
- [Background] Hayashi M, Wilson NH. Failure risk of posterior composites with post-operative sensitivity. Oper Dent. 2003 Nov-Dec;28(6):681-8. PMID 14653280
- [Background] Kaurani M, Bhagwat SV. Clinical evaluation of postoperative sensitivity in composite resin restorations using various liners. N Y State Dent J. 2007 Mar;73(2):23-9. PMID 17472181
- [Background] Letzel H. Survival rates and reasons for failure of posterior composite restorations in multicentre clinical trial. J Dent. 1989;17 Suppl 1:S10-7; discussion S26-8. doi: 10.1016/0300-5712(89)90156-5. PMID 2659634
- [Background] Liang K-Y, Zeger SL (1986). Longitudinal data analysis using generalized linear models. Biometrika 73:13-22.
- [Background] Lundin SA, Rasmusson CG. Clinical evaluation of a resin composite and bonding agent in Class I and II restorations: 2-year results. Quintessence Int. 2004 Oct;35(9):758-62. PMID 15471000
- [Background] Miguez PA, Pereira PN, Foxton RM, Walter R, Nunes MF, Swift EJ Jr. Effects of flowable resin on bond strength and gap formation in Class I restorations. Dent Mater. 2004 Nov;20(9):839-45. doi: 10.1016/j.dental.2003.10.015. PMID 15451239
- [Background] Ommerborn MA, Schneider C, Giraki M, Schafer R, Singh P, Franz M, Raab WH. In vivo evaluation of noncarious cervical lesions in sleep bruxism subjects. J Prosthet Dent. 2007 Aug;98(2):150-8. doi: 10.1016/S0022-3913(07)60048-1. PMID 17692596
- [Background] Opdam NJ, Feilzer AJ, Roeters JJ, Smale I. Class I occlusal composite resin restorations: in vivo post-operative sensitivity, wall adaptation, and microleakage. Am J Dent. 1998 Oct;11(5):229-34. PMID 10388382
- [Background] Perdigao J, Geraldeli S, Hodges JS. Total-etch versus self-etch adhesive: effect on postoperative sensitivity. J Am Dent Assoc. 2003 Dec;134(12):1621-9. doi: 10.14219/jada.archive.2003.0109. PMID 14719760
- [Background] Perdigao J, Anauate-Netto C, Carmo AR, Hodges JS, Cordeiro HJ, Lewgoy HR, Dutra-Correa M, Castilhos N, Amore R. The effect of adhesive and flowable composite on postoperative sensitivity: 2-week results. Quintessence Int. 2004 Nov-Dec;35(10):777-84. PMID 15553285
- [Background] Perdigao J, Dutra-Correa M, Castilhos N, Carmo AR, Anauate-Netto C, Cordeiro HJ, Amore R, Lewgoy HR. One-year clinical performance of self-etch adhesives in posterior restorations. Am J Dent. 2007 Apr;20(2):125-33. PMID 17542208
- [Background] Perdigao J, Dutra-Correa M, Anauate-Netto C, Castilhos N, Carmo AR, Lewgoy HR, Amore R, Cordeiro HJ. Two-year clinical evaluation of self-etching adhesives in posterior restorations. J Adhes Dent. 2009 Apr;11(2):149-59. PMID 19492717
- [Background] Rosin M, Steffen H, Konschake C, Greese U, Teichmann D, Hartmann A, Meyer G. One-year evaluation of an Ormocer restorative-a multipractice clinical trial. Clin Oral Investig. 2003 Mar;7(1):20-6. doi: 10.1007/s00784-002-0189-9. Epub 2003 Feb 4. PMID 12673433
- [Background] Sadeghi M, Lynch CD, Shahamat N. Eighteen-month clinical evaluation of microhybrid, packable and nanofilled resin composites in Class I restorations. J Oral Rehabil. 2010 Jul;37(7):532-7. doi: 10.1111/j.1365-2842.2010.02073.x. Epub 2010 Feb 25. PMID 20202097
- [Background] Sobral MA, Garone-Netto N, Luz MA, Santos AP. Prevention of postoperative tooth sensitivity: a preliminary clinical trial. J Oral Rehabil. 2005 Sep;32(9):661-8. doi: 10.1111/j.1365-2842.2005.01479.x. PMID 16102079
- [Background] Swift EJ Jr, Ritter AV, Heymann HO, Sturdevant JR, Wilder AD Jr. 36-month clinical evaluation of two adhesives and microhybrid resin composites in Class I restorations. Am J Dent. 2008 Jun;21(3):148-52. PMID 18686764
- [Background] Turkun LS, Turkun M, Ozata F. Clinical performance of a packable resin composite for a period of 3 years. Quintessence Int. 2005 May;36(5):365-72. PMID 15892534
- [Background] van Dijken JW, Sunnegardh-Gronberg K. A two-year clinical evaluation of a new calcium aluminate cement in Class II cavities. Acta Odontol Scand. 2003 Aug;61(4):235-40. doi: 10.1080/00016350310004575. PMID 14582592
- [Background] Wegehaupt F, Betke H, Solloch N, Musch U, Wiegand A, Attin T. Influence of cavity lining and remaining dentin thickness on the occurrence of postoperative hypersensitivity of composite restorations. J Adhes Dent. 2009 Apr;11(2):137-41. PMID 19492715
- [Background] Wilson NH, Wilson MA, Smith GA. A clinical trial of a new visible light-cured composite restorative-- initial findings and one-year results. Quintessence Int. 1985 Apr;16(4):281-90. No abstract available. PMID 3859888
- [Background] Yip KH, Poon BK, Chu FC, Poon EC, Kong FY, Smales RJ. Clinical evaluation of packable and conventional hybrid resin-based composites for posterior restorations in permanent teeth: results at 12 months. J Am Dent Assoc. 2003 Dec;134(12):1581-9. doi: 10.14219/jada.archive.2003.0103. PMID 14719754
- [Background] Johansson A, Haraldson T, Omar R, Kiliaridis S, Carlsson GE. A system for assessing the severity and progression of occlusal tooth wear. J Oral Rehabil. 1993 Mar;20(2):125-31. doi: 10.1111/j.1365-2842.1993.tb01596.x. PMID 8468624
- [Background] Lavigne GJ, Manzini C, Kato T (2005). Sleep Bruxism. In: Principles and practice of sleep medicine. MH Kryger, T Roth and WC Dement editors. Philadelphia: Elsevier, pp. 946-59
- [Derived] Curro FA, Vena D, Naftolin F, Terracio L, Thompson VP. The PBRN initiative: transforming new technologies to improve patient care. J Dent Res. 2012 Jul;91(7 Suppl):12S-20S. doi: 10.1177/0022034512447948. PMID 22699662